CLINICAL TRIAL: NCT05095961
Title: Effect of Pre-operative Oral Steroids on Blood Loss in Endoscopic Sinus Surgery for Chronic Rhinosinusitis Without Polyps
Brief Title: Pre-operative Steroids in CRSsP
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Technical difficulties encountered with recording intraoperative blood loss; unable to proceed with study.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5210327
Record Dates: First submitted 2021-09-29; First posted 2021-10-27 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Chronic Sinus Disease; Chronic Sinusitis, Ethmoidal; Chronic Sinusitis, Sphenoidal; Chronic Sinusitis - Maxillary Bilateral; Chronic Sinusitis - Frontoethmoidal
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Patient's will be randomized to one of two groups: pre-operative oral steroids or no control
Who Masked: Outcomes Assessor
Masking Description: Clinicians grading blood loss and surgical field disability on the recorded video footage will be blinded to patient identity and group status. Data analysis will be done by a blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pre-operative oral steroids (Experimental): Patients will be given a course of oral prednisone (30mg daily) for 5 days.
  Interventions: Drug: Prednisone
- Control (No Intervention): No pre-operative medication will be prescribed

INTERVENTIONS:
Drug: Prednisone — 5 day course of oral prednisone pre-operatively. 30mg per day.
  Arms: Pre-operative oral steroids

SUMMARY:
Randomized controlled trial to determine the effectiveness of a five-day course of pre-operative oral steroids on decreasing intra-operative blood loss during endoscopic sinus surgery.

DETAILED DESCRIPTION:
The study will be a randomized cohort study, and patients will be recruited before surgery. Following randomization, patients will be given either a course of Prednisone (30 milligrams per day for 5 days, to be started five days prior to surgery) or no additional pre-operative prescriptions besides what is clinically determined by their treating physician. Patients will be scheduled for surgery and undergo functional endoscopic sinus surgery with timing as clinically indicated.

During endoscopic sinus surgery, surgical video will be recorded and stored on encrypted, flash drives with unique, non PHI, indicators to identify drives. Subsequently, each video will be graded by two, blinded surgeons for field visualization and thoroughness of dissection. Intra-operative blood loss will also be recorded. Post-operative data through 30 days post-operatively will be collected including: post-operative complications, resolution of symptoms, and nasal crusting during post-operative follow up. Following completion of data collection, these data will be analyzed by a separate, blinded investigator.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between the ages of 18 and 99 years of age with a diagnosis of chronic rhinosinusitis without polyps who are being scheduled for functional endoscopic sinus surgery

Exclusion Criteria:

* Patients under 18 years old, patients with a condition in which the use of systemic corticosteroids is contraindicated (poorly controlled diabetes mellitus, poorly controlled hypertension, active or untreated tuberculosis, active viral or fungal infection, acute angle glaucoma, osteoporosis, or acute congestive heart failure) patients allergic to corticosteroids, or, patients unwilling or unable to take the prescribed course of pre-operative steroids.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Intra-operative blood loss - 1 | Intra-operative
  Measured intra-operative blood loss (in milliliters) as assessed by standard measure (total of blood in the suction canister [less the irrigation used])
Intra-operative blood loss - 2 | Intra-operative
  Blinded assessors grading of blood loss (in milliliters) as assessed by standard measure (total of blood in the suction canister [less the irrigation used])
Surgical field visibility | Intra-operative
  Blinded assessor's grading of surgical field visualization

SECONDARY OUTCOMES:
Patient intolerance of steroids | Pre-operative
  Patient report of intolerable adverse effects of pre-operative steroids

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Chan, MD, Principal Investigator — Loma Linda University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Govindaraj S, Adappa ND, Kennedy DW. Endoscopic sinus surgery: evolution and technical innovations. J Laryngol Otol. 2010 Mar;124(3):242-50. doi: 10.1017/S0022215109991368. Epub 2009 Nov 23. PMID 19930748
- [Background] Linder TE, Simmen D, Stool SE. Revolutionary inventions in the 20th century. The history of endoscopy. Arch Otolaryngol Head Neck Surg. 1997 Nov;123(11):1161-3. doi: 10.1001/archotol.1997.01900110011001. PMID 9366694
- [Background] Moffatt DC, McQuitty RA, Wright AE, Kamucheka TS, Haider AL, Chaaban MR. Evaluating the Role of Anesthesia on Intraoperative Blood Loss and Visibility during Endoscopic Sinus Surgery: A Meta-analysis. Am J Rhinol Allergy. 2021 Sep;35(5):674-684. doi: 10.1177/1945892421989155. Epub 2021 Jan 21. PMID 33478255
- [Background] Wawrzyniak K, Burduk PK, Cywinski JB, Kusza K, Kazmierczak W. Improved quality of surgical field during endoscopic sinus surgery after clonidine premedication--a pilot study. Int Forum Allergy Rhinol. 2014 Jul;4(7):542-7. doi: 10.1002/alr.21308. Epub 2014 Mar 3. PMID 24591266
- [Background] Sieskiewicz A, Olszewska E, Rogowski M, Grycz E. Preoperative corticosteroid oral therapy and intraoperative bleeding during functional endoscopic sinus surgery in patients with severe nasal polyposis: a preliminary investigation. Ann Otol Rhinol Laryngol. 2006 Jul;115(7):490-4. doi: 10.1177/000348940611500702. PMID 16900802
- [Background] Gunel C, Basak HS, Bleier BS. Oral steroids and intraoperative bleeding during endoscopic sinus surgery. B-ENT. 2015;11(2):123-8. PMID 26563012
- [Background] Hwang SH, Seo JH, Joo YH, Kang JM. Does the Preoperative Administration of Steroids Reduce Intraoperative Bleeding during Endoscopic Surgery of Nasal Polyps? Otolaryngol Head Neck Surg. 2016 Dec;155(6):949-955. doi: 10.1177/0194599816663455. Epub 2016 Aug 23. PMID 27554509